CLINICAL TRIAL: NCT02163174
Title: Pentoxifylline Therapy of Late-onset Sepsis in Preterm Infants: A Randomized Controlled Trial.
Brief Title: Pentoxifylline and Late Onset Sepsis in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abd Elazeez Attala Shabaan (Other)
Responsible Party: Sponsor-Investigator, Abd Elazeez Attala Shabaan, Associate Professor of Pediatrics, Mansoura faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12345; R88 (Other: local institutional research board)
Record Dates: First submitted 2014-06-06; First posted 2014-06-13 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Neonatal Late Onset Sepsis
Keywords: neonatal; pentoxifylline; randomized controlled trial
MeSH Terms: conditions — Neonatal Sepsis | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentoxyfilline arm (Active Comparator): Pentoxifylline 5 mg/kg/hr for 6 hours on 6 successive days in addition to antibiotics.
  Interventions: Drug: Pentoxifylline (PTX)
- Placebo arm (Placebo Comparator): Intravenous saline as a Placebo 5 mg/kg/hr for 6 hours on 6 successive days in addition to antibiotics.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline (PTX) — Patients were randomly assigned to receive intravenous Pentoxifylline 5 mg/kg/hr for 6 hours on 6 successive days in addition to antibiotics
  Other Names: Trental (brand name)
  Arms: Pentoxyfilline arm
Drug: Placebo — Patients were randomly assigned to receive intravenous normal saline 5 mg/kg/hr for 6 hours on 6 successive days as a placebo in addition to antibiotics.
  Arms: Placebo arm

SUMMARY:
* Hypothesis: The investigators hypothesized that Pentoxifylline has potent anti-inflammatory effect which can augment the antimicrobial effect of antibiotics in treatment of Late onset sepsis (LOS) in preterm infants thus decreasing neonatal mortality and morbidity.
* The purpose of this study: to assess the efficacy and safety of Pentoxifylline as an adjunct to antibiotic therapy on mortality and morbidity of preterm infants with LOS.

DETAILED DESCRIPTION:
* Role of pentoxifylline, a phosphodiesterase inhibitor, in reducing mortality associated with neonatal sepsis is not well studied.
* Hypothesis: we hypothesized that Pentoxifylline has potent anti-inflammatory effect which can augment the antimicrobial effect of antibiotics in treatment of Late onset sepsis (LOS) in preterm infants thus decreasing neonatal mortality and morbidity.
* Purpose of the study: to assess the efficacy and safety of Pentoxifylline as an adjunct to antibiotic therapy on mortality and morbidity of preterm infants with LOS.
* Design: A prospective, randomized, double-blind clinical trial.
* Setting: Neonatal Intensive Care Unit, Mansoura University Children's Hospital.
* Patients: 120 preterm infants with suspected or confirmed LOS.
* Intervention: Enrolled infants were randomly assigned to receive intravenous Pentoxifylline (5 mg/kg/hr for 6 hours on 6 successive days) or placebo in addition to antibiotics.
* Primary outcome: Death before hospital discharge.
* Secondary outcomes: Length of hospital stay, duration of respiratory support, duration of antibiotics use, chronic lung disease, necrotizing enterocolitis, intraventricular hemorrhage, periventricular leukomalacia, retinopathy of prematurity, Serum levels of Tumor necrosis factor, C-Reactive protein levels, and adverse effects of Pentoxifylline.

ELIGIBILITY:
Inclusion Criteria:

- Appropriate for gestational age preterm infants with suspected or confirmed late onset sepsis

Exclusion Criteria:

* Preterm infants with major congenital malformations
* Preterm infants with chromosomal anomalies
* Preterm infants with inborn-errors of metabolism
* Preterm infants with congenital infection

Ages: 5 Days to 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality | Expected 10 weeks postnatal age
  Mortality before discharge from neonatal intensive care unit

SECONDARY OUTCOMES:
Length of hospital stay | Expected average of 8 weeks post natal age
  Duration of hospital admission (days)
Duration of respiratory support | Expected 4 to 6 weeks postnatal age
  Duration of respiratory support including oxygen, Continuous Positive Airway Pressure, mechanical ventilation(days)
Duration of antibiotics use | Expected 3 to 5 weeks postnatal age
  Duration of treatment of sepsis including meningitis
Chronic lung disease | By 36 weeks corrected gestational age
  Need for oxygen by 36 weeks corrected gestational age
Necrotising enterocolitis | Expected 6 weeks
  Bell clinical and radiological criteria
Intraventricular haemorrhage | Expected 2 weeks
  By cranial ultrasound grading
Periventricular leukomalacia | Expected 8 weeks
  By cranial ultrasound
Retinopathy of prematurity | Expected 8 weeks
  Ophthalmologist using Ret-Cam
Serum levels of Tumor necrosis factor-α, C-Reactive protein | 6 days after intervention
Adverse effects of Pentoxifylline | Up to 10 days after intervention
  Adverse effects of Pentoxifylline such as feeding intolerance, thrombocytopenia and cholestasis.

CONTACTS AND LOCATIONS:
Overall Officials: Abd Elazeez AT Shabaan, PhD, Principal Investigator — Mansoura University, Faculty of Medicine
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, Eldakahlia, Egypt

REFERENCES:
- [Derived] Shabaan AE, Nasef N, Shouman B, Nour I, Mesbah A, Abdel-Hady H. Pentoxifylline therapy for late-onset sepsis in preterm infants: a randomized controlled trial. Pediatr Infect Dis J. 2015 Jun;34(6):e143-8. doi: 10.1097/INF.0000000000000698. PMID 25970116